CLINICAL TRIAL: NCT01237587
Title: Effect of Duloxetine 30/60 mg Once Daily Versus Placebo in Adolescents With Juvenile Primary Fibromyalgia Syndrome
Brief Title: A Study of Duloxetine in Adolescents With Juvenile Primary Fibromyalgia Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14099; F1J-MC-HMGW (Other: Eli Lilly and Company); CTRI/2011/07/001866 (Registry Identifier: Clinical Trials Registry India)
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Fibromyalgia
Keywords: Adolescents; Juvenile Primary Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): Blinded treatment period: 30mg or 60mg once daily for 13 weeks
  Open label extension: 30mg or 60mg Duloxetine once daily for 26 weeks
  Taper period: 30mg Duloxetine or placebo once daily for 1 week.
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Blinded treatment period:Placebo once daily for 13 weeks
  Open label extension: 30mg or 60mg Duloxetine once daily for 26 weeks
  Taper period: 30mg Duloxetine or placebo once daily for 1 week.
  Interventions: Drug: Duloxetine; Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Administered orally
  Other Names: LY248686
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether duloxetine is safe and effective in the treatment of adolescents with Juvenile Primary Fibromyalgia Syndrome (JPFS).

This trial consists of two distinct study periods. A blinded treatment period of 13 weeks and an open label extension period of 26 weeks.

ELIGIBILITY:
Inclusion Criteria

* Meet criteria for primary JPFS
* Have a score of greater than or equal to 4 on Brief Pain Inventory (BPI) average pain severity (Item 3) during screening
* Female participants must have a negative serum pregnancy test during screening
* Participant's parent/legal representative and participant judged to be reliable to keep all appointments for clinical tests and procedures
* Participant's parent/legal representative and participant must have a degree of understanding such that they can communicate intelligently
* Participants must be capable of swallowing investigational product whole
* Participants must have venous access sufficient to allow blood sampling and be compliant with blood draws

Exclusion Criteria:

* Currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device or concurrently enrolled in any other type of medical research
* Previously completed or withdrawn after randomization from a study investigating duloxetine
* Known hypersensitivity to duloxetine or any of the inactive ingredients, or have frequent or severe allergic reactions to multiple medications
* Treated with duloxetine within the last 6 months. Will not likely benefit from duloxetine treatment, in the opinion of the investigator or have had prior nonresponse or inadequate tolerance to duloxetine
* Pain symptoms related to traumatic injury, past surgery, structural bone or joint disease or regional pain syndrome that will interfere with interpretation of outcome measures
* Currently have evidence of rheumatologic disorder or have a current diagnosis of rheumatoid arthritis, inflammatory arthritis, or infectious arthritis, or an autoimmune disease (for example, systemic lupus erythematosus)
* Have a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) Axis I condition, currently or within the past year, except major depressive disorder (MDD) and/or generalized anxiety disorder (GAD), adjustment disorder or specific phobias with primary investigator approval
* Have a current secondary DSM-IV Axis I condition of attention-deficit/hyperactivity disorder that requires pharmacologic treatment
* Lifetime DSM-IV Axis I diagnosis of psychosis, bipolar disorder, or schizoaffective disorder
* DSM-IV Axis II disorder which would interfere with protocol compliance
* History of substance abuse or dependence within the 6 months
* Positive urine drug screen for any substances of abuse or excluded medication
* Family history of 1 or more first-degree relatives with diagnosed bipolar I disorder
* Significant suicide attempt within 1 year of screening or are currently at suicidal risk in the opinion of the investigator
* Weight less than 20 kilogram (kg) at screening
* History of seizure disorder (other than febrile seizures)
* Taking any excluded medications that cannot be discontinued at screening
* Fluoxetine within 30 days prior to completion of screening
* Monoamine oxidase inhibitor (MAOI) within 14 days of screening; or the potential need to use an MAOI during the study or within 5 days of discontinuation of investigational product
* Abnormal thyroid-stimulating hormone (TSH) concentrations
* Uncontrolled narrow-angle glaucoma
* Acute liver injury (such as hepatitis) or severe cirrhosis (Child-Pugh Class C)
* Serious or unstable medical illness
* Female participants who are either pregnant, nursing or have recently given birth

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2011-03; Primary Completion 2017-05-31 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 : Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (33):
- United States (26):
  - NoesisPharma, Phoenix, Arizona
  - Loma Linda University School of Medicine, Loma Linda, California
  - Synergy Clinical Research, National City, California
  - Connecticut Clinical Trials LLC, Cromwell, Connecticut
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - Palm Beach Research Center, West Palm Beach, Florida
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Riley Hosptial for Children, Indianapolis, Indiana
  - Kentucky Medical Research Center, Lexington, Kentucky
  - Mercy Health Research, St Louis, Missouri
  - Healthy Perspectives Innovative Mental Health Services, PL, Nashua, New Hampshire
  - Albuquerque Neurosciences, Albuquerque, New Mexico
  - Bioscience Research, LLC, Mount Kisco, New York
  - Richmond Behavorial Associates, Staten Island, New York
  - Neurobehavioral Clinical Research, Canton, Ohio
  - Univ of Cincinnati College of Medicine, Cincinnati, Ohio
  - North Star Research, Middleburg Heights, Ohio
  - Neuropsychiatric Center, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - CRI Lifetree, Philadelphia, Pennsylvania
  - Holston Medical Group Clinical Research, Kingsport, Tennessee
  - Arthritis and Osteoporosis Center of South Texas, San Antonio, Texas
  - Bateman Horne Center of Excellence, Salt Lake City, Utah
  - NeuroScience, Inc., Herndon, Virginia
  - Advanced Pain Management, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán, Argentina
- India (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mysore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raipur
- Puerto Rico (2):
  - Centro de Investigaciones Clinicas, San Juan
  - Centro Pediatrico Paseos, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Upadhyaya HP, Arnold LM, Alaka K, Qiao M, Williams D, Mehta R. Efficacy and safety of duloxetine versus placebo in adolescents with juvenile fibromyalgia: results from a randomized controlled trial. Pediatr Rheumatol Online J. 2019 May 28;17(1):27. doi: 10.1186/s12969-019-0325-6. PMID 31138224
- See also: Click here for more information about this study: A Study of Duloxetine in Adolescents With Juvenile Primary Fibromyalgia Syndrome — http://www.lillytrialguide.com/en-US/studies/fibromyalgia/HMGW#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 week Double-Blind Treatment Phase (Acute Phase), followed by 26 week Open-Label Extension Treatment Phase (Extension Phase), followed by 1 week Taper/Discontinuation Phase.
Groups:
- Duloxetine/Duloxetine: Participants received flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 13 weeks during double blind treatment period (Acute Phase) and flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 26 weeks during open label extension treatment period (Extension Phase).
  Participants who received higher doses of Duloxetine in acute & extension phase received gradually lower doses of duloxetine & participants on lower doses of Duloxetine in acute phase received placebo during 1-week tapering phase.
- Placebo/Duloxetine: Participants received Placebo orally once daily (QD) for 13 weeks during double blind treatment phase and flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 26 weeks during open label extension treatment period (Extension Phase).
  Participants who received placebo in acute phase received placebo & participants who received higher doses of Duloxetine in extension phase received gradually lower doses of duloxetine during1-week tapering phase.
Period: Double Blind Treatment (Acute Phase)
Arm/Group | Duloxetine/Duloxetine | Placebo/Duloxetine
Started | 91 | 93
Received at Least One Dose of Study Drug | 91 | 93
Completed | 74 | 75
Not Completed | 17 | 18
Not completed — Adverse Event | 5 | 1
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — Parent/Caregiver Decision | 2 | 4
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal by Subject | 3 | 4
Period: Open Label Treatment (Extension Phase)
Arm/Group | Duloxetine/Duloxetine | Placebo/Duloxetine
Started | 74 | 75
Received at Least One Dose of Study Drug | 74 | 75
Completed | 56 | 50
Not Completed | 18 | 25
Not completed — Lost to Follow-up | 4 | 3
Not completed — Adverse Event | 5 | 5
Not completed — Lack of Efficacy | 2 | 4
Not completed — Parent/Guardian Decision | 2 | 4
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Sponsor Decision | 1 | 0
Not completed — Physician Decision | 4 | 4
Period: Taper Phase
Arm/Group | Duloxetine/Duloxetine | Placebo/Duloxetine
Started | 36 (Participants who discontinued Acute or Extension phase had an option to enter tapering phase.) | 44 (Participants who discontinued Acute or Extension phase had an option to enter tapering phase.)
Completed | 31 | 34
Not Completed | 5 | 10
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Lack of Efficacy | 2 | 5
Not completed — Parent/Guardian Decision | 0 | 2
Not completed — Sponsor Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Duloxetine: Participants received flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 13 weeks during double blind treatment period (Acute Phase) and flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 26 weeks during open label extension treatment period (Extension Phase).
  Participants who received higher doses of Duloxetine in acute & extension phase received gradually lower doses of duloxetine & participants on lower doses of Duloxetine in acute phase received placebo during 1-week tapering phase.
- Placebo: Participants received Placebo orally once daily (QD) for 13 weeks during double blind treatment phase and flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 26 weeks during open label extension treatment period (Extension Phase).
  Participants who received placebo in acute phase received placebo & participants who received higher doses of Duloxetine in extension phase received gradually lower doses of duloxetine during 1-week tapering phase.
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 91 | 93 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.74 (1.379) | 15.33 (1.421) | 15.53 (1.411)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 65 | 138
  Male | 18 | 28 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 39 | 75
  Not Hispanic or Latino | 54 | 54 | 108
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 8 | 15
  White | 72 | 70 | 142
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 2 | 3 | 5
  Argentina | 19 | 19 | 38
  United States | 64 | 64 | 128
  India | 6 | 7 | 13
Brief Pain Inventory (BPI) Modified short form (SF) Adolescent version (AV) [Mean (Standard Deviation); unit: units on a scale] — BPI Modified SF AV is a scale that measures severity & interference of pain. Severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine). 4 questions assessing severity for worst pain, least pain, average pain in past 24 hours, & pain right now.Interference scores range from 0 (does not interfere) to 10 (completely interferes).7 questions assessing interference of pain in past 24 hours on general activity, mood, walking ability, normal work, relations with other people, sleep, & enjoyment of life. Adolescent Version has 8th question for interference of pain on school work. Population: All randomized participants who had baseline BPI score.
  units on a scale
    Average Pain: number analyzed (Participants) | 90 | 91 | 181
    Average Pain | 5.7 (1.37) | 5.6 (1.55) | 5.65 (1.46)
    Worst Pain | 7.1 (1.8) | 6.9 (1.9) | 7.0 (1.9)
    Least Pain | 3.7 (2.1) | 3.8 (2.0) | 3.8 (2.1)
    Pain Right Now | 5.2 (2.4) | 5.2 (2.3) | 5.2 (2.4)
    General Activity | 5.2 (2.0) | 5.1 (2.0) | 5.2 (2.3)
    Mood | 4.9 (2.6) | 5.0 (2.6) | 5.0 (2.6)
    Walking Ability | 4.1 (2.8) | 4.5 (2.8) | 4.3 (2.8)
    Normal Work | 4.6 (2.6) | 4.9 (2.5) | 4.8 (2.6)
    Relations with other people | 3.7 (2.7) | 3.7 (2.8) | 3.7 (2.8)
    Sleep | 5.9 (2.8) | 5.5 (3.0) | 5.7 (2.9)
    Enjoyment of Life | 4.1 (3.1) | 4.3 (2.8) | 4.2 (3.0)
    School Work | 4.8 (3.0) | 4.3 (3.2) | 4.6 (3.1)
Pediatric Pain Questionnaire (PPQ) [Mean (Standard Deviation); unit: mm] — Pediatric Pain Questionnaire (PPQ) is a self-reported scale that measures the severity for "pain now," worst pain, and average pain in the past week with 100 millimeter (mm) VAS (Visual Analog Scale). The severity scores range from 0 (no hurting, no discomfort, no pain) to 100 (hurting a whole lot, very uncomfortable, severe pain). Population: All randomized participants who had baseline PPQ score.
  mm
    Average Pain: number analyzed (Participants) | 87 | 86 | 173
    Average Pain | 61.8 (19.5) | 58.1 (22.3) | 58.94 (20.9)
    Worst Pain: number analyzed (Participants) | 87 | 86 | 173
    Worst Pain | 77.4 (20.3) | 75.5 (20.4) | 76.5 (20.4)
    pain now: number analyzed (Participants) | 87 | 86 | 173
    pain now | 50.1 (27.5) | 52.0 (25.2) | 51.0 (26.4)
Clinical Global Impression (CGI) Severity: Mental Illness [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression of Severity: Mental Illness (CGI-S: Mental Illness) scale evaluates the severity of any diagnosed, comorbid Axis I/II condition. The scoring ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Participants without a diagnosed Axis I/II condition should receive a score of 1 (normal, not at all ill). Population: All randomized participants who had baseline CGI mental illness score.
  units on a scale
    number analyzed (Participants) | 90 | 92 | 182
    (all) | 2.1 (1.2) | 2.0 (1.1) | 2.05 (1.15)
Clinical Global Impression (CGI) Severity: Overall Illness [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression of Severity: Overall Illness (CGI-S: Overall Illness) scale evaluates the severity of the overall illness of Juvenile Primary Fibromyalgia Syndrome (JPFS), including all relevant, associated symptoms. The scoring ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The scoring is based on observed and reported symptoms and behaviors over the past 7 days that are ongoing at the time of the Study Visit. Population: All randomized participants who had baseline CGI overall illness score.
  units on a scale
    number analyzed (Participants) | 90 | 92 | 182
    (all) | 4.1 (0.9) | 4.1 (0.8) | 4.1 (0.9)
Functional Disability Inventory (FDI) Child score [Mean (Standard Deviation); unit: units on a scale] — Functional Disability Inventory-child form (FDI-child) is a self-reported scale to assess the physical trouble or difficulty the child has doing regular activities. This scale contains 15 items. Each item is scored on a 0- to-4-point scale (0 = no trouble, 1 = a little trouble, 2 = some trouble, 3 = a lot of trouble, 4 = impossible).The total score ranges from 0 to 60. The higher the score, the more physical trouble or difficulty the child has doing regular activities. Population: All randomized participants who had baseline FDI child score.
  units on a scale
    number analyzed (Participants) | 87 | 88 | 175
    (all) | 23.3 (11.1) | 22.3 (9.9) | 22.8 (10.5)
Functional Disability Inventory (FDI) Parent Score [Mean (Standard Deviation); unit: units on a scale] — Functional Disability Inventory-parent form (FDI-parent) contains the same items as FDI-child, but is reported by parent/legal representative. The total score range from 0 to 60. The higher the score, the more physical trouble or difficulty the child has doing regular activities. Population: All randomized participants who had baseline FDI parent score.
  units on a scale
    number analyzed (Participants) | 86 | 87 | 173
    (all) | 22.4 (11.4) | 22.3 (10.7) | 22.4 (11.1)
Children's Depression Inventory (CDI) [Mean (Standard Deviation); unit: units on a scale] — Children's Depression Inventory (CDI) is modeled after the Beck Depression Inventory and is a 27-item self-reported, symptom-oriented scale designed for school aged children and adolescents. Each item is scored on a 0-to-2-point scale (in increasing severity) and thus the total score ranges from 0 to 54. The higher the score, the more severe the depression. Population: All randomized participants who had baseline CDI score.
  units on a scale
    number analyzed (Participants) | 89 | 89 | 178
    (all) | 13.5 (7.1) | 13.1 (7.7) | 13.3 (7.4)
Multidimensional Anxiety Scale for Children (MASC) [Mean (Standard Deviation); unit: units on a scale] — MASC consists of 39 items that comprise 4 factors. Each item is scored on a 0 to 3-point scale (0-never to 3-often).
  1. Physical symptoms (tense/restless and somatic/autonomic) - 12 items with score range 0 to 36.
  2. Social anxiety (humiliation/rejection and public performance fears) - 9 items with score range of 0 to 27.
  3. Harm avoidance (perfectionism and anxious coping) - 9 items with score range of 0 to 27.
  4. Separation anxiety - 9 items with score range of 0 to 27. Total score ranges from 0 to 117. Higher the total score, the more severe the anxiety. Population: All randomized participants who had baseline MASC score.
  units on a scale
    Physical Symptoms: number analyzed (Participants) | 89 | 89 | 178
    Physical Symptoms | 13.6 (7.3) | 13.6 (7.6) | 13.6 (7.5)
    Harm Avoidance: number analyzed (Participants) | 89 | 89 | 178
    Harm Avoidance | 15.0 (4.2) | 14.4 (4.7) | 14.7 (4.5)
    Social Anxiety: number analyzed (Participants) | 89 | 89 | 178
    Social Anxiety | 9.8 (6.3) | 9.8 (6.3) | 9.8 (6.6)
    Separation/Panic: number analyzed (Participants) | 89 | 89 | 178
    Separation/Panic | 6.7 (4.9) | 6.0 (4.5) | 6.4 (4.7)
    Total Score: number analyzed (Participants) | 89 | 89 | 178
    Total Score | 45.1 (16.6) | 43.9 (18.7) | 44.5 (17.65)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory (BPI) Modified Short Form-adolescent Version 24 Hour Average Pain Severity Item
Description: Brief Pain Inventory (BPI) modified short form is a self-reported scale that measures the severity of pain and the interference of pain on function, Severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine). Severity of pain is measured based on the average pain experienced over the past 24-hours.
  Mixed Model Repeated Measure (MMRM) model with terms for treatment, pooled investigator, visit, baseline, treatment by visit, and baseline by visit was used to produce Least Square (LS) means.
Time Frame: Baseline, 13 weeks
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline BPI average pain score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine - Acute: Participants received 30 or 60 mg Duloxetine orally once daily (QD) for 13 weeks.
- Placebo - Acute: Participants received Placebo orally once daily (QD) for 13 weeks.
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 76 | 76
units on a scale | -1.62 (0.247) | -0.97 (0.244)
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Test type: Superiority; p = 0.052, Repeated Measures; LS mean change difference = -0.65, 95% CI 2-sided [-1.30 to 0.00], Standard Error of Mean 0.330

2. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Brief Pain Inventory (BPI) Modified Short Form-Adolescent Version Severity and Interference Items
Description: The Brief Pain Inventory (BPI) - Modified Short Form Adolescent Version is a self-reported scale that measures the severity of pain and the interference of pain on function. The Severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine).There are 4 questions assessing the severity for worst pain, least pain, average pain in the past 24 hours (which is the primary efficacy measure), and the pain right now. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 original questions assessing the interference of pain in the past 24 hours on the following: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The BPI: Adolescent Version added an eighth interference question to assess interference of pain on school work.
  MMRM model with terms for treatment, pooled investigator, visit, baseline, treatment by visit, and baseline by visit was used to produce LS means.
Time Frame: Baseline, 13 weeks
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline BPI severity & interferences items score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 76 | 76
units on a scale
  Worst Pain | -1.58 (0.270) | -0.90 (0.266)
  Least Pain | -1.08 (0.239) | -0.47 (0.236)
  Pain Right Now | -1.56 (0.274) | -1.05 (0.271)
  General Activity | -2.00 (0.262) | -1.03 (0.258)
  Mood | -2.00 (0.269) | -1.46 (0.265)
  Walking ability | -1.30 (0.266) | -1.09 (0.262)
  Normal Work | -1.49 (0.277) | -1.21 (0.274)
  Relations With Other People | -1.87 (0.237) | -1.07 (0.233)
  Sleep | -1.40 (0.343) | -1.05 (0.338)
  Enjoyment of Life | -1.76 (0.253) | -1.47 (0.250)
  School Work | -1.68 (0.316) | -1.08 (0.313)
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Worst Pain; Test type: Superiority; p = .059, Mixed Models Analysis; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.40 to 0.03], Standard Error of Mean 0.360
Statistical Analysis 2: Comparison: Duloxetine - Acute vs Placebo - Acute; Least Pain; Test type: Superiority; p = 0.059, Mixed Models Analysis; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-1.24 to 0.02], Standard Error of Mean 0.319
Statistical Analysis 3: Comparison: Duloxetine - Acute vs Placebo - Acute; Pain Right Now; Test type: Superiority; p = .165, Mixed Models Analysis; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.23 to 0.21], Standard Error of Mean 0.365
Statistical Analysis 4: Comparison: Duloxetine - Acute vs Placebo - Acute; General Activity; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.65 to -0.30], Standard Error of Mean 0.344
Statistical Analysis 5: Comparison: Duloxetine - Acute vs Placebo - Acute; Mood; Test type: Superiority; p = .128, Mixed Models Analysis; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-1.25 to 0.16], Standard Error of Mean 0.356
Statistical Analysis 6: Comparison: Duloxetine - Acute vs Placebo - Acute; Walking ability; Test type: Superiority; p = .560, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.90 to 0.49], Standard Error of Mean 0.352
Statistical Analysis 7: Comparison: Duloxetine - Acute vs Placebo - Acute; Normal Work; Test type: Superiority; p = 0.448, Mixed Models Analysis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.01 to 0.45], Standard Error of Mean 0.371
Statistical Analysis 8: Comparison: Duloxetine - Acute vs Placebo - Acute; Relations With Other; Test type: Superiority; p = .011, Mixed Models Analysis; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.42 to -0.19], Standard Error of Mean 0.312
Statistical Analysis 9: Comparison: Duloxetine - Acute vs Placebo - Acute; Sleep; Test type: Superiority; p = .443, Mixed Models Analysis; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.25 to 0.55], Standard Error of Mean 0.454
Statistical Analysis 10: Comparison: Duloxetine - Acute vs Placebo - Acute; Enjoyment of Life; Test type: Superiority; p = .390, Mixed Models Analysis; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.96 to 0.38], Standard Error of Mean 0.338
Statistical Analysis 11: Comparison: Duloxetine - Acute vs Placebo - Acute; School Work; Test type: Superiority; p = .160, Mixed Models Analysis; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-1.44 to 0.24], Standard Error of Mean 0.424

3. Secondary Outcome: Maintenance Effect in Acute Phase Responders on the Brief Pain Inventory (BPI) Modified Short Form-adolescent Version 24 Hour Average Pain Severity Item
Description: Brief Pain Inventory (BPI) modified short form is a self-reported scale that measures the severity of pain and the interference of pain on function.Severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine). Severity of pain is measured based on the average pain experienced over the past 24-hours.
  Acute phase responders: Participants with ≥30% pain reduction from baseline on the BPI average pain severity measure at the last non-missing assessment in acute phase.
Time Frame: Baseline (Extension Phase), 39 weeks
Population: All randomized participants in duloxetine only arm with ≥30% pain reduction from baseline on the BPI average pain severity measure at the last non-missing assessment in acute phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duloxetine/Duloxetine - Extension: Participants received flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 13 weeks during double blind treatment period (Acute Phase) and flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 26 weeks during open label extension treatment phase.
Arm/Group | Duloxetine/Duloxetine - Extension
Number analyzed (Participants) | 44
units on a scale | -3.4 (1.24)

4. Secondary Outcome: Number of Participants With Greater Than or Equal to 30% Reduction From Baseline in BPI 24 Hour Average Pain Severity Score at 13 Weeks
Description: Brief Pain Inventory (BPI) modified short form is a self-reported scale that measures the severity of pain and interference of pain on function, Severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine). Severity of pain is measured based on the average pain experienced over the past 24-hours.
  Percent reduction of BPI 24 hour average pain from baseline to last observation carried forward (LOCF).
Time Frame: 13 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 90 | 91
Participants | 47 | 33
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Test type: Superiority; p = .051, Fisher Exact

5. Secondary Outcome: Number of Participants With Greater Than or Equal to 50% Reduction From Baseline in BPI 24 Hour Average Pain Severity Score at 13 Weeks
Description: as for outcome 4
Time Frame: 13 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 90 | 91
Participants | 36 | 22
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Test type: Superiority; p = .038, Fisher Exact

6. Secondary Outcome: Change From Baseline in Pediatric Pain Questionnaire (PPQ) Item Scores
Description: Pediatric Pain Questionnaire (PPQ) is a self-reported scale that measures the severity for "pain now," worst pain, and average pain in the past week with 100 mm VAS (Visual Analog Scale). The severity scores range from 0 (no hurting, no discomfort, no pain) to 100 (hurting a whole lot, very uncomfortable, severe pain).
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for treatment, pooled investigator and baseline value.
Time Frame: Baseline, 13 weeks
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline PPQ score.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 87 | 86
mm
  Average Pain Score | -11.03 (2.982) | -9.41 (2.946)
  Worst Pain Score | -14.36 (3.367) | -8.46 (3.322)
  Pain Score Right Now | -8.99 (3.092) | -7.20 (3.065)
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Average Pain Score; Test type: Superiority; p = .669, ANCOVA; Mean Difference (Final Values) = 1.62, 95% CI 2-sided [-9.10 to 5.86]
Statistical Analysis 2: Comparison: Duloxetine - Acute vs Placebo - Acute; Worst Pain Score; Test type: Superiority; p = .169, ANCOVA; Mean Difference (Final Values) = -5.90, 95% CI 2-sided [-14.32 to 2.53]
Statistical Analysis 3: Comparison: Duloxetine - Acute vs Placebo - Acute; Pain Score Right Now; Test type: Superiority; p = .647, ANCOVA; Mean Difference (Final Values) = -1.79, 95% CI 2-sided [-9.53 to 5.94]

7. Secondary Outcome: Change From Baseline in Clinical Global Impression (CGI) Severity: Overall Illness Score
Description: Clinical Global Impression of Severity: Overall Illness (CGI-S: Overall Illness) scale evaluates the severity of the overall illness of JPFS, including all relevant, associated symptoms. The scoring ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The scoring is based on observed and reported symptoms and behaviors over the past 7 days that are ongoing at the time of the Study Visit.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS mean with terms for treatment, pooled investigator and baseline value.
Time Frame: Baseline, 13 weeks
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline CGI-S overall illness score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 90 | 92
units on a scale | -0.88 (0.121) | -0.66 (0.118)
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Test type: Superiority; p = .146, ANCOVA; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.52 to 0.08]

8. Secondary Outcome: Change From Baseline in Clinical Global Impression (CGI) Severity: Mental Illness Score
Description: Clinical Global Impression of Severity: Mental Illness (CGI-S: Mental Illness) scale evaluates the severity of any diagnosed, comorbid Axis I/II condition. The scoring ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Participants without a diagnosed Axis I/II condition should receive a score of 1 (normal, not at all ill).
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS mean with terms for treatment, pooled investigator and baseline value.
Time Frame: Baseline, 13 weeks
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline CGI-S mental illness score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 90 | 92
units on a scale | -0.16 (0.089) | -0.15 (0.087)
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Test type: Superiority; p = .927, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.23 to 0.21]

9. Secondary Outcome: Change From Baseline in Functional Disability Inventory Child Form (FDI-Child)
Description: Functional Disability Inventory-child form (FDI-child) is a self-reported scale to assess the physical trouble or difficulty the child has doing regular activities. This scale contains 15 items. Each item is scored on a 0- to-4-point scale (0 = no trouble, 1 = a little trouble, 2 = some trouble, 3 = a lot of trouble, 4 = impossible).The total score ranges from 0 to 60. The higher the score, the more physical trouble or difficulty the child has doing regular activities.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for treatment, pooled investigator and baseline value.
Time Frame: Baseline, 13 weeks
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline FDI child scale score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 87 | 88
units on a scale | -3.97 (1.038) | -5.00 (1.021)
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Test type: Superiority; p = .431, ANCOVA; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [-1.54 to 3.59]

10. Secondary Outcome: Change From Baseline in Functional Disability Inventory Parent Form (FDI-Parent)
Description: Functional Disability Inventory-parent form (FDI-parent) contains the same items as FDI-child, but is reported by parent/legal representative. The total score range from 0 to 60. The higher the score, the more physical trouble or difficulty the child has doing regular activities.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for treatment, pooled investigator and baseline value.
Time Frame: Baseline, 13 weeks
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline FDI-parent scale score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 86 | 87
units on a scale | -3.25 (1.152) | -4.17 (1.139)
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Test type: Superiority; p = .529, ANCOVA; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [-1.95 to 3.79]

11. Secondary Outcome: Change From Baseline in Children's Depression Inventory (CDI)
Description: Children's Depression Inventory (CDI) is modeled after the Beck Depression Inventory and is a 27-item self-reported, symptom-oriented scale designed for school-aged children and adolescents. Each item is scored on a 0-to-2-point scale (in increasing severity) and thus the total score ranges from 0 to 54. The higher the score, the more severe the depression.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for treatment, pooled investigator and baseline value.
Time Frame: Baseline, 13 weeks
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline CDI score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 89 | 89
units on a scale | -3.28 (0.682) | -2.45 (0.674)
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Test type: Superiority; p = .335, ANCOVA; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-2.52 to 0.86]

12. Secondary Outcome: Change From Baseline in Multidimensional Anxiety Scale for Children (MASC)
Description: Multidimensional Anxiety Scale for Children (MASC) is a self-reported scale developed to assess anxiety in children and adolescents. The MASC consists of 39 items that comprise 4 factors with each item scored on a 0-to-3-point scale (0-never true about me, 1-rarely true about me, 2- sometimes true about me, 3-often true about me). : 1) physical symptoms (tense/restless and somatic/autonomic)-12 items with score range 0 to 36; 2) social anxiety (humiliation/rejection and public performance fears)-9 items with score range of 0 to 27; 3) harm avoidance (perfectionism and anxious coping)-9 items with score range of 0 to 27; and 4) separation anxiety-9 items with score range of 0 to 27. Total score ranges from 0 to 117. The higher the total score, the more severe the anxiety.Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for treatment, pooled investigator and baseline value.
Time Frame: Baseline, 13 weeks
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline MASC score.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for treatment, pooled investigator and baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine - Acute | Placebo - Acute
Number analyzed (Participants) | 89 | 89
units on a scale
  Physical Symptoms | -1.39 (0.663) | -1.44 (0.652)
  Harm Avoidance | -1.34 (0.507) | -0.78 (0.501)
  Social Anxiety | -1.86 (0.497) | -1.42 (0.489)
  Separation/Panic | -1.62 (0.393) | -1.43 (0.389)
  Total Score | -6.21 (1.575) | -4.99 (1.558)
Statistical Analysis 1: Comparison: Duloxetine - Acute vs Placebo - Acute; Physical Symptoms Score; Test type: Superiority; p = .955, ANCOVA; Mean Difference (Final Values) = .05, 95% CI 2-sided [-1.59 to 1.68]
Statistical Analysis 2: Comparison: Duloxetine - Acute vs Placebo - Acute; Harm Avoidance; Test type: Superiority; p = .381, ANCOVA; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.82 to 0.70]
Statistical Analysis 3: Comparison: Duloxetine - Acute vs Placebo - Acute; Social Anxiety; Test type: Superiority; p = .486, ANCOVA; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.66 to 0.79]
Statistical Analysis 4: Comparison: Duloxetine - Acute vs Placebo - Acute; Separation/Panic; Test type: Superiority; p = .700, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-1.17 to 0.79]
Statistical Analysis 5: Comparison: Duloxetine - Acute vs Placebo - Acute; Total Score; Test type: Superiority; p = .540, ANCOVA; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-5.12 to 2.69]

13. Secondary Outcome: Change From Baseline to 39 Week Endpoint in Brief Pain Inventory (BPI) Modified Short Form-adolescent Version Severity and Interference Items
Description: The BPI - Modified Short Form Adolescent Version is a self-reported scale that measures the severity of pain and the interference of pain on function. The Severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine).There are 4 questions assessing the severity for worst pain, least pain, average pain in the past 24 hours (which is the primary efficacy measure), and the pain right now. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 original questions assessing the interference of pain in the past 24 hours on the following: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The BPI: Adolescent Version added an eighth interference question to assess interference of pain on school work.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for pooled investigator and baseline value.
Time Frame: Baseline (extension phase), 39 weeks
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post baseline BPI severity & interferences items scores.
  Baseline for extension phase is defined as the last non-missing value in acute phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine/Duloxetine - Extension Phase: Participants received flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 13 weeks during double blind treatment period (Acute Phase) and flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 26 weeks during open label extension treatment period (Extension Phase).
- Placebo/Duloxetine - Extension Phase: Participants received Placebo orally once daily (QD) for 13 weeks during double blind treatment phase and flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 26 weeks during open label extension treatment period (Extension Phase).
Arm/Group | Duloxetine/Duloxetine - Extension Phase | Placebo/Duloxetine - Extension Phase
Number analyzed (Participants) | 74 | 75
units on a scale
  Worst Pain | -0.65 (0.262) | -0.80 (0.256)
  Least Pain | -0.29 (0.218) | -0.45 (0.212)
  Pain Right Now | -0.38 (0.259) | -0.29 (0.252)
  General Activity | -0.18 (0.233) | 0.20 (0.229)
  Mood | -0.15 (0.270) | -0.25 (0.258)
  Walking Ability | -0.24 (0.260) | -0.21 (0.253)
  Normal Work | -0.62 (0.231) | -0.32 (0.226)
  Relations with Other People | -0.12 (0.229) | -0.41 (0.222)
  Sleep | -0.63 (0.292) | -0.54 (0.284)
  Enjoyment of Life | -0.25 (0.243) | -0.26 (0.236)
  School Work | -0.59 (0.278) | -0.06 (0.271)

14. Secondary Outcome: Change From Baseline in Pediatric Pain Questionnaire (PPQ) Item Scores
Description: Pediatric Pain Questionnaire (PPQ) is a self-reported scale that measures the severity for "pain now," worst pain, and average pain in the past week with 100 mm VAS (Visual Analog Scale). The severity scores range from 0 (no hurting, no discomfort, no pain) to 100 (hurting a whole lot, very uncomfortable, severe pain).
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for pooled investigator and baseline value.
Time Frame: Baseline (extension phase), 39 weeks
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post baseline PPQ measurement.
  Baseline for extension phase is defined as the last non-missing value in acute phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine - Extension Phase | Placebo/Duloxetine - Extension Phase
Number analyzed (Participants) | 68 | 60
units on a scale
  Average Pain Score | -10.65 (3.080) | -6.44 (3.296)
  Worst Pain Score | -4.15 (3.127) | -8.06 (3.677)
  Score Right Now | -4.74 (3.075) | -6.34 (3.335)

15. Secondary Outcome: Change From Baseline in Clinical Global Impression (CGI) Severity: Overall Illness Score
Description: Clinical Global Impression of Severity: Overall Illness (CGI-S: Overall Illness) scale evaluates the severity of the overall illness of JPFS, including all relevant, associated symptoms. The scoring ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The scoring is based on observed and reported symptoms and behaviors over the past 7 days that are ongoing at the time of the Study Visit.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS mean with terms for pooled investigator and baseline value.
Time Frame: Baseline (extension phase), 39 weeks
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post baseline CGI overall illness measurement.
  Baseline for extension phase is defined as the last non-missing value in acute phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine - Extension Phase | Placebo/Duloxetine - Extension Phase
Number analyzed (Participants) | 74 | 75
units on a scale | -0.67 (0.125) | -0.67 (0.121)

16. Secondary Outcome: Change From Baseline in Clinical Global Impression (CGI) Severity: Mental Illness Score
Description: Clinical Global Impression of Severity: Mental Illness (CGI-S: Mental Illness) scale evaluates the severity of any diagnosed, comorbid Axis I/II condition. The scoring ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Participants without a diagnosed Axis I/II condition should receive a score of 1 (normal, not at all ill).
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS mean with terms for pooled investigator and baseline value.
Time Frame: Baseline (extension phase), 39 weeks
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post baseline CGI mental Illness measurement.
  Baseline for extension phase is defined as the last non-missing value in acute phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine - Extension Phase | Placebo/Duloxetine - Extension Phase
Number analyzed (Participants) | 74 | 75
units on a scale | -0.20 (0.104) | -0.24 (0.101)

17. Secondary Outcome: Change From Baseline in Functional Disability Inventory Child Form (FDI-child)
Description: Functional Disability Inventory-child form (FDI-child) is a self-reported scale to assess the physical trouble or difficulty the child has doing regular activities. This scale contains 15 items. Each item is scored on a 0- to-4-point scale (0 = no trouble, 1 = a little trouble, 2 = some trouble, 3 = a lot of trouble, 4 = impossible).The total score ranges from 0 to 60. The higher the score, the more physical trouble or difficulty the child has doing regular activities.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for pooled investigator and baseline value.
Time Frame: Baseline (extension phase), 39 weeks
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post baseline FDI-child measurement.
  Baseline for extension phase is defined as the last non-missing value in acute phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine - Extension Phase | Placebo/Duloxetine - Extension Phase
Number analyzed (Participants) | 67 | 62
units on a scale | -1.71 (1.202) | -1.03 (1.267)

18. Secondary Outcome: Change From Baseline in Functional Disability Inventory Parent Form (FDI-parent)
Description: Functional Disability Inventory-parent form (FDI-parent) contains the same items as FDI-child, but is reported by parent/legal representative. The total score range from 0 to 60. The higher the score, the more physical trouble or difficulty the child has doing regular activities.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for pooled investigator and baseline value.
Time Frame: Baseline (extension phase), 39 weeks
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post baseline FDI-parent measurement.
  Baseline for extension phase is defined as the last non-missing value in acute phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine - Extension Phase | Placebo/Duloxetine - Extension Phase
Number analyzed (Participants) | 68 | 60
units on a scale | -3.49 (1.227) | -2.27 (1.327)

19. Secondary Outcome: Change From Baseline in Children's Depression Inventory (CDI)
Description: Children's Depression Inventory (CDI) is modeled after the Beck Depression Inventory and is a 27-item self-reported, symptom-oriented scale designed for school-aged children and adolescents. Each item is scored on a 0-to-2-point scale (in increasing severity) and thus the total score ranges from 0 to 54. The higher the score, the more severe the depression.
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) was used to produce LS means with terms for pooled investigator and baseline value.
Time Frame: Baseline (extension phase), 39 weeks
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post baseline CDI measurement.
  Baseline for extension phase is defined as the last non-missing value in acute phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine - Extension Phase | Placebo/Duloxetine - Extension Phase
Number analyzed (Participants) | 74 | 74
units on a scale | -0.42 (0.703) | -1.41 (0.681)

20. Secondary Outcome: Change From Baseline in Multidimensional Anxiety Scale for Children (MASC)
Description: Multidimensional Anxiety Scale for Children (MASC) is a self-reported scale developed to assess anxiety in children and adolescents. The MASC consists of 39 items that comprise 4 factors with each item scored on a 0-to-3-point scale (0-never true about me, 1-rarely true about me, 2- sometimes true about me, 3-often true about me). : 1) physical symptoms (tense/restless and somatic/autonomic)-12 items with score range 0 to 36; 2) social anxiety (humiliation/rejection and public performance fears)-9 items with score range of 0 to 27; 3) harm avoidance (perfectionism and anxious coping)-9 items with score range of 0 to 27; and 4) separation anxiety-9 items with score range of 0 to 27. Total score ranges from 0 to 117. The higher the total score, the more severe the anxiety.ANCOVA model with last observation carried forward (LOCF) was used to produce LS means with terms for pooled investigator and baseline value.
Time Frame: Baseline (extension phase), 39 weeks
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post baseline MASC measurement.
  Baseline for extension phase is defined as the last non-missing value in acute phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine - Extension Phase | Placebo/Duloxetine - Extension Phase
Number analyzed (Participants) | 74 | 74
units on a scale
  Physical Symptoms | -0.63 (0.715) | -0.92 (0.692)
  Harm Avoidance | 0.23 (0.485) | 0.10 (0.471)
  Social Anxiety | -0.11 (0.487) | -0.02 (0.472)
  Separation/Panic | -0.06 (0.371) | 0.01 (0.361)
  Total Score | -0.55 (1.478) | -0.78 (1.432)

ADVERSE EVENTS:
Time Frame: up to 39 weeks
Groups:
- Duloxetine - Acute: Participants received 30 or 60 mg Duloxetine orally once daily (QD) for 13 weeks during Acute phase.
- Placebo - Acute: Participants received Placebo orally once daily (QD) for 13 weeks during Acute phase.
- Duloxetine/Duloxetine - Extension: Participants received flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 13 weeks during double blind treatment period (Acute Phase) and flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 26 weeks during open label extension treatment period (Extension Phase).
- Placebo/Duloxetine - Extension: Participants received Placebo orally once daily (QD) for 13 weeks during double blind treatment phase and flexible doses of 30 or 60 milligram (mg) Duloxetine orally once daily (QD) for 26 weeks during open label extension treatment period (Extension Phase).
- Duloxetine 60/Duloxetine 30 - Taper: Participants who received 60mg Duloxetine in acute & extension phase received 30mg of Duloxetine in taper phase.
- Placebo/Placebo - Taper: Participants who received placebo or 30mg Duloxetine in acute phase received placebo in Taper phase.
Arm/Group | Duloxetine - Acute | Placebo - Acute | Duloxetine/Duloxetine - Extension | Placebo/Duloxetine - Extension | Duloxetine 60/Duloxetine 30 - Taper | Placebo/Placebo - Taper
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/93 | 0/74 | 0/75 | 0/77 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/91 | 0/93 | 3/74 | 3/75 | 0/77 | 0/3
Other Adverse Events (participants affected / at risk) | 74/91 | 58/93 | 52/74 | 54/75 | 7/77 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine - Acute (N=91) | Placebo - Acute (N=93) | Duloxetine/Duloxetine - Extension (N=74) | Placebo/Duloxetine - Extension (N=75) | Duloxetine 60/Duloxetine 30 - Taper (N=77) | Placebo/Placebo - Taper (N=3)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Duloxetine - Acute (N=91) | Placebo - Acute (N=93) | Duloxetine/Duloxetine - Extension (N=74) | Placebo/Duloxetine - Extension (N=75) | Duloxetine 60/Duloxetine 30 - Taper (N=77) | Placebo/Placebo - Taper (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2) | 6 (8) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 23 (30) | 14 (16) | 10 (14) | 22 (26) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (19) | 5 (5) | 4 (4) | 8 (9) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 5 (6) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (11) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2) | 6 (6) | 4 (4) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 14 (14) | 3 (5) | 6 (6) | 8 (9) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 8 (10) | 9 (13) | 4 (4) | 3 (4) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 13 (15) | 10 (14) | 6 (8) | 5 (9) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 8 (8) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2/73 (2) | 4/65 (6) | 2/61 (2) | 2/53 (5) | 0/60 (0) | 0/2 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/18 (0) | 0/28 (0) | 1/13 (1) | 0/22 (0) | 0/17 (0) | 0/1 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (4):
  • Study Protocol: Protocol (2010-10-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT01237587/Prot_000.pdf
  • Study Protocol: Protocol Amendment (a) (2011-07-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT01237587/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT01237587/SAP_002.pdf
  • Study Protocol: Protocol Amendment (b) (2013-04-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT01237587/Prot_003.pdf